CLINICAL TRIAL: NCT00620594
Title: A Phase I/II, Multi-center, Open-label Study of BEZ235, Administered Orally on a Continuous Daily Dosing Schedule in Adult Patients With Advanced Solid Malignancies Including Patients With Advanced Breast Cancer
Brief Title: A Phase I/II Study of BEZ235 in Patients With Advanced Solid Malignancies Enriched by Patients With Advanced Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBEZ235A2101; 2006-004353-23 (EudraCT Number)
Record Dates: First submitted 2008-02-08; First posted 2008-02-21 (Estimated); Last update posted 2020-12-09 (Actual); Status verified 2017-02

CONDITIONS: Breast Cancer; Advanced Solid Tumors; Cowden Syndrome
Keywords: Neoplasms; breast neoplasms; breast diseases; solid tumors; BEZ235; breast cancer; PI3K Inhibitor; Phosphatidylinositol 3; kinase; advanced
MeSH Terms: conditions — Breast Neoplasms; Hamartoma Syndrome, Multiple; Neoplasms; Breast Diseases | interventions — dactolisib

ARMS (4):
- BEZ235 Alone, Dose Escalation (Experimental)
  Interventions: Drug: BEZ235
- BEZ235 + trastuzumab, Dose Escalation (Experimental)
  Interventions: Drug: BEZ235
- BEZ235 Alone, MTD Expansion (Experimental)
  Interventions: Drug: BEZ235
- BEZ235 + Trastuzumab, MTD Expansion (Experimental)
  Interventions: Drug: BEZ235

INTERVENTIONS:
Drug: BEZ235

SUMMARY:
This is a first-in-human, phase I/Ib clinical research study with BEZ235, an inhibitor of phosphatidylinositol 3'-kinase (PI3K). The study consists of a dose escalation part followed by a safety dose expansion part:

Dose escalation part (advanced solid tumors, including patients with breast cancer being treated with trastuzumab):

Patients receive oral BEZ235 once daily on days 1-28 of the first course. Courses will repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of at least 3 patients receive escalating doses of BEZ235, as single agent or in combination with trastuzumab, until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose expected to produce during the first course of treatment dose-limiting toxicity in 33% of patients.

Once the MTD has been defined, the safety expansion parts of the trial will be opened for enrollment.

Safety dose expansion part (advanced solid tumors, including patients with breast cancer being treated with trastuzumab):

Patients will be treated with BEZ235, as single agent or in combination with trastuzumab, given at the MTD, once daily. Treatment of patients will continue until disease progression or occurrence of unacceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

[Single agent dose escalation arm]: Patients with histologically-confirmed, advanced unresectable solid tumors including CS patients who have progressed on (or not been able to tolerate) standard therapy within three months before screening visit or for whom no standard anticancer therapy exists.

[Combination part]: Patients with metastatic HER2+ Breast Cancer, after failure of trastuzumab treatment. Eligible patients will have to have tumors carrying molecular alterations of PIK3CA and/or PTEN.

[Single agent safety expansion arm]: Patients with histologically-confirmed, advanced unresectable solid tumors including CS patients who have progressed on (or not been able to tolerate) standard therapy within three months before screening visit or for whom no standard anticancer therapy exists. Patients will be prescreened for molecular alterations affecting PIK3CA and/or PTEN. Patients with NSCLC will also be pre-screened for EGFR mutation.

Exclusion Criteria:

* Patients who have brain metastases, which are progressive and/or requiring medical intervention for symptom control
* Prior treatment with a PI3K inhibitor
* Acute or chronic liver disease or renal disease
* Acute or chronic pancreatitis
* Patients with unresolved diarrhea ≥ CTCAE grade 2
* Impaired cardiac function or clinically significant cardiac diseases
* Patients with diabetes mellitus requiring insulin treatment
* Patients with known coagulopathies
* Patients with a history of photosensitivity reactions to other drugs
* Any of the following ophthalmological findings:
* Progressive eye disease that could lead to severe loss of visual acuity or visual field
* loss during the study period
* Inability to perform the ophthalmic procedures required in this protocol
* Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g. active or uncontrolled infection) that could cause unacceptable safety risks or compromise compliance with the protocol.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2006-12-21 (Actual); Primary Completion 2013-01-08 (Actual); Study Completion 2013-01-08 (Actual)

PRIMARY OUTCOMES:
determine the maximum Tolerated Dose (MTD) of BEZ235 as single agent and in combination with trastuzumab (Dose escalation part) | at end of study
assess the safety & tolerability of BEZ235 SDS as single agent and in combination with trastuzumab administered to patients at the MTD level (Safety expansion part) | at end of study

SECONDARY OUTCOMES:
assess the safety and tolerability of the various formulations of BEZ235 | at end of study
Asses the Pharmacokinetics of BEZ235 which includes AUC, Cmax, Tmax, t1/2 as endpoints | at end of study
Preliminary anti-tumor activity (tumor response) of BEZ235 SDS as single agent and in combination with trastuzumab | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (14):
- United States (9):
  - University of California at Los Angeles JonssonComprehensiveCancerCtr, Los Angeles, California
  - Yale University School of Medicine YaleCancerCtr-ClinTrialsOffice, New Haven, Connecticut
  - Dana Farber Cancer Institute Clinical Trials ProjectManager, Boston, Massachusetts
  - Nevada Cancer Institute NVCC - Huntsman, Las Vegas, Nevada
  - Cancer Centers of the Carolinas CCC Faris, Greenville, South Carolina
  - Sarah Cannon Research Institute Dept.ofSarahCannonCancerCtr(2), Nashville, Tennessee
  - Baylor Health Care System/Sammons Cancer Center Baylor- Sammons, Dallas, Texas
  - University of Texas/MD Anderson Cancer Center Thoractic Head/Neck Med.Onc(2), Houston, Texas
  - Tyler Cancer Center TCC, Tyler, Texas
- Novartis Investigative Site, Essen, Germany
- Novartis Investigative Site, Amsterdam, Netherlands
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Valencia, Valencia
- Novartis Investigative Site, Manchester, United Kingdom

REFERENCES:
- See also: Results for CBEZ235A2101 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=10543